CLINICAL TRIAL: NCT05964478
Title: Hands4Health: Hand Hygiene, Water Quality and Sanitation in Schools Not Connected to a Functional Water Supply System: a Cluster-randomized Controlled Trial in Nigeria and Palestine
Brief Title: Hands4Health: A Multi-component Intervention on Hand Hygiene & Well-being in Schools in Nigeria & Palestine (H4H)
Acronym: H4H
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Tropical & Public Health Institute (Other)
Collaborators: University of Applied Sciences and Arts Northwestern Switzerland (Other); Terre des Hommes (Unknown); CESVI (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 7F-l 0345.03.01A
Record Dates: First submitted 2023-07-19; First posted 2023-07-28 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Hand Hygiene; Handwashing Behaviour; Well-Being
Keywords: Behaviour Change; WASH Infrastructure; Handwashing Station; Handwashing; Students; Primary Schools; Humanitarian

STUDY DESIGN:
Intervention Model Description: The study is a multi-center Cluster Randomised Controlled Trial being conducted across two countries. Within each country, there will be two arms: an intervention arm and a control arm.
  The intervention arm will receive a comprehensive multi-component intervention package. On the other hand, the control arm will not receive the intervention package during the data collection phase, serving as a comparison group.
  However, It will receive the same intervention package (with potential improvements) once the data collection period concludes, specifically at the endline assessment after one year from the baseline
Masking Description: The laboratory technicians involved in the processing and analysis of the hand rinse samples will be masked and therefore do not know if the sample comes from the intervention or the control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm of schools in Nigeria and Palestine (Experimental): The participating schools in this arm will receive the multi-component hand hygiene intervention package for a duration of one year
  Interventions: Other: Multi-component hand hygiene intervention in primary schools not connected to functional water supply system in Nigeria and Palestine
- Control arm of schools in Nigeria and Palestine (No Intervention): The participating schools in this arm will not receive the multi-component hand hygiene intervention package until the conclusion of the study, which occurs one year after the completion of data collection at the endline assessment

INTERVENTIONS:
Other: Multi-component hand hygiene intervention in primary schools not connected to functional water supply system in Nigeria and Palestine — Each participating school receives: (i) Two Gravit'eau handwashing stations (http://www.graviteau.ch): these systems recycle on-site greywater and operate through gravity and a manual foot pump, and can be produced locally. (ii) Behavior change activities: Developed by a group of expert psychologists (http://www.ranasmosler.com/ranas), utilizing the risks, attitudes, norms, abilities, and self-regulation (RANAS) approach. (iii) WASH infrastructure rehabilitation and soap dispenser installation. (iv) Controlled chlorine monitoring: Equipment provided for monitoring chlorine concentration in water storage, with staff training. (v) Preventive maintenance: Trained circuit rider inspects infrastructure regularly under WASH committee supervision
  Other Names: Gravit'eau handwashing system; RANAS4schools; Chlorination support; Preventive maintenance
  Arms: Intervention arm of schools in Nigeria and Palestine

SUMMARY:
The aim of this study is to assess the impact of the hands4health hand hygiene multi-component intervention on students and teachers in primary schools with limited access to water in Nigeria and Palestine. To evaluate the effects of the intervention, the investigators will involve the participants in the included schools in the following data collection methods, including (i) a survey regarding their thoughts, behaviours, and practices related to handwashing at school, (ii) structured observation of their handwashing behaviour (iii) hand rinse sample collection to check for bacteria on their hands, (iv) absenteeism tracking through a daily journal to record the reasons for any absences, with a specific focus on identifying if they are related to hygiene-related diseases, and (v) discussions and interviews to gather their perspectives on the perceived impacts of the intervention on their health and well-being.

The investigators will collect data using these methods before the intervention starts, a few months after it begins, and again one year later. The schools will be randomly divided into two groups: one group will receive the intervention activities, including handwashing station/rehabilitation of water, sanitation and hygiene infrastructure, behavioural change intervention, capacity development, and management support. The other group will not receive any intervention until the end of the study. By comparing the two groups, the investigators will determine if the intervention had any impact on health determinants including, hygiene infrastructure, handwashing knowledge, behaviour, beliefs, etc.

DETAILED DESCRIPTION:
The overall project will follow a multi-center cluster-randomized controlled trial (cRCT) design. Prior to this study, a group of schools in the study's target areas were surveyed by the Tdh (in Nigeria) and Cesvi (in Palestine) using the Facility Evaluation Tool for WASH in Schools (FACET WINS) which is a monitoring tool for WASH delivery services in schools. From these schools a subsample was identified which fulfils certain inclusion criteria (see Eligibility). This subsample was handed over to the local Tdh and Cesvi collaborators who carefully assessed the security situation around the schools. The Tdh and Cesvi collaborators then selected 26 facilities per country, which are most probable to still be accessible for data collection within the next year. These 26 schools will then be allocated to the two arms (intervention vs. control) with covariate constrained stratified randomization using computer-generated randomization code provided by a statistician not involved in any field activities. The intervention arm will receive the full intervention package (see multi-component intervention in primary schools). The control arm will receive nothing for the duration of the intervention (12 months). Afterwards, they will receive the same intervention package with potential improvements identified in the former intervention group.

Objectives of the study:

* Primary objective: Evaluate the effects of the H4H multi-component intervention on hand hygiene of primary school students in Nigeria and Palestine.
* Secondary objectives:

  * Evaluate the effects of the H4H multi-component on the well-being of primary school students in Nigeria and Palestine
  * Assess the effect of the H4H multi-component package on hygiene-related risks, attitudes, norms, abilities and self-regulation (RANAS) behavioural factors of primary school students
  * Explore the associations of personal, physical and social contextual factors with hand hygiene and the well-being of primary school students in Palestine
  * Explore the perceived impacts of the H4H multi-component package on the health and well-being of primary school students
* Explorative object: Assess the effect of the H4H multi-component package on hygiene-related health outcomes and absenteeism incidence of primary school students in Nigeria and Palestine.

In the schools, the investigators selected 50 eligible students from each school from one or two classes within the age group of 10-12 years using random sampling. If a school had a single class consisting of ≥ 50 students within the study's target age group, the investigators selected the sample from that class. However, if no class with the target age group had more than 50 students, the investigators randomly selected two classes from within the target age group and selected the sample from these classes. For different data collection modules, the investigators randomly selected subsets from the 50 previously selected students.

The modules of the study incudes qualitative and quantitative data approaches in order to enable a triangulation of the overall project results. The following modules will be used in the cRCT and the overall project: (i) Module 1: Combined RANAS and well-being survey, (ii) Module 2: Structured handwashing observations, (iii) Module 3: Microbiological analysis of hand rinse samples, (iv) Module 4: Diary approach for health outcomes and absenteeism, (v) Module 5: personal, physical and social contextual factors survey (vi) Module 6: Focus Group Discussions (FGDs) and (vii) Module 7: Key informant interviews (KIIs)..

Local collaborators from Tdh and Cesvi and the regional Ministries of Education (MoE) were involved from the study's kick-off meeting onwards and are regularly being consulted in bi-weekly meetings and additional ToC workshops led by Skat Foundation. The data collection methods for each module will be described in further detail:

(i) Module 1: Combined RANAS and well-being survey: The survey will be developed through RANAS approach that targets the underlying psychological factors that are postulated as important precursors for effective behaviour change by the model. These factors include handwashing-related perceived risks, attitudes, norms, abilities and self-regulation. The well-being of the participants will be assessed in the survey using the KINDL tool which is designed to measure health-related quality of life in children and adolescents by looking into different domains of well-being (e.g. physical, mental and school). The survey will also contain questions assessing the perceived sufficiency and safety of the water supply, satisfaction with the available infrastructure for handwashing, and obstacles to water access. The survey will be administered to a randomly selected subset of 25 students per primary school three times in total; as a baseline survey before the implementation of the intervention package, about three months after the intervention and about a year after the baseline survey with the software Open Data Kit (ODK) Central (version 2022.3.1) on Android tablets. Informed consent forms will be obtained from the participants' guardians before the day of data collection. In addition, oral assent will also be obtained from the participants at the beginning of the interview for filling out the survey.

(ii) Module 2: Structured handwashing observations: The observations will be administered three times at the same time points as the survey in Module 1. To be able to assess individual behaviours and link them to data collected using other tools, all of the students in the classes selected for the study will be assigned coloured badges with their unique IDs. Students will be informed that they are randomly assigned the colours. However, the data collector will agree with the school teachers on a specific colour to be assigned to the 50 students selected for the study from these classes. The observation will start at 9:00 am (60 minutes before the breakfast break) and end at 12:00 pm (90 minutes after the break). The data collector will pilot the observation process before the intervention and in coordination with the school staff.

The occurrence of handwashing with soap will be observed for each of the two critical handwashing events (after using the toilet and before eating) for each included student. To observe handwashing before eating (study's primary outcome), the investigators will engage participants in a painting activity, followed by a popcorn snack, which should prompt handwashing. During snack time, observers stationed at handwashing points will document who washes their hands. Observations will also include other handwashing opportunities, such as after toilet use. Outcomes will indicate whether or not handwashing with soap occurred at these key events, with some considerations for unforeseen field complications. If feasible, the investigators will observe the handwashing steps of students who do wash their hands. Consent for observation will be obtained at a school level, from the principal of the school, as well as from the parents.

(iii) Module 3: Microbiological analysis of hand rinse samples: This module focuses on the microbiological analysis of hand rinse samples from a random subset of 12 students three times at the same time points as the survey in Module 1 and observation in Module 2. The modified glove juice method is the process used for that and it involves shaking and massaging participant's hands in 350 mL of clean water contained in a 710 mL Whirl-Pak bag (NASCO Corp., Fort Atkinson, WI), followed by drying. The bags with samples are kept on ice and processed within four hours. Using membrane filtration, the investigators will detect E. Coli and total coliforms colony-forming units (CFUs). This will involve filtering the bag contents through a 47-mm-diameter 0.45 µm cellulose filter, applying the filter to growth media, and incubating it at 35°C ± 0.5°C for a duration of 24 hours. the investigators plan to filter 100 mL per bag; however, the exact amount of mL will be established during piloting as the volume used is dependent on the degree of bacterial contamination on the hands. The investigators will utilize compact dry plates to detect E.coli and total coliforms, and the detection limits will be calculated based on the filtrate volume and Whirl-Pak volume. The lower detection limit of CFUs will be calculated by dividing 1 CFU/plate by the filtrate volume and then multiplying it with the total Whirl-Pak volume of 350 mL. The upper detection limit will be calculated by dividing 500 CFUs/plate by the filtrate volume and then multiplying it with the Whirl-Pak volume. For analysis, CFUs per hand will be normalized and log10 transformed.

(iv) Module 4: Diary approach for health outcomes and absenteeism incidence: The approach uses a diary method to track hygiene-related health outcomes and absenteeism post-intervention. The key measure is hygiene-related absenteeism, tied to conditions like diarrhea, respiratory and skin infections, helminth infections, head lice, and trachoma. A teacher in each school will record daily absences and reasons in an electronic/paper diary. To account for the cluster design, the investigators will separately calculate hygiene-related absenteeism rates for each medical condition in each school by dividing the number of absences by student-weeks, yielding rates per 100 student-weeks.

(v) Module 5: personal, physical and social contextual factors survey. The cultural and contextual factors that may influence students' handwashing and well-being will be covered in this survey. Given the unique stressors of military occupation in Palestine, it's crucial to understand these conditions' impact on life beyond school. The investigators will analyse determinants of hygiene behaviour before starting the intervention, providing insight into how to maximize effectiveness for broader hygiene interventions in Palestine. The study uses a cross-sectional baseline design, with an initial assessment conducted before school randomization. Parents of the 50 included students will complete a survey assessing household hygiene services, their hygiene knowledge and habits, and their child's hygiene behaviour.

(vi) Module 6: Focus Group Discussions (FGDs): The FGDs generate extensive data quicker than individual interviews. The investigators will conduct 10 gender-separated FGDs in the selected schools during autumn 2023. This separation also encourages open, free-speaking environments without fear of teasing or embarrassment. Each group will consist of 5-8 students, ensuring a fair representation from each class participating in the study. To avoid dominance issues, the investigators will ensure all students within a group are of the same age. Furthermore, there will be 5 FGDs specifically designed for 5-8 teachers from schools involved in the intervention. The team conducting the FGDs, ideally including the SwissTPH PhD student, will consist of a moderator and a note-taker. FGDs will be tape-recorded, transcribed, and translated into English for analysis, with observations noted in a field research journal. Analysis will be conducted using MaxQDA (VERBI Software, Marburg, Germany) or NVivo software (QSR International, Melbourne, Australia).

(vii) Module 7: Key informant interviews (KIIs): The key informant interviews will be with education ministry stakeholders, school committee members, and community leaders, to gain detailed insights into specific issues and proposed solutions. This data will be collected in autumn 2023, providing depth that FGDs might miss due to group dynamics. Interviewers, trained similarly to those for FGDs, will audio record interviews, with transcripts translated into English for analysis using either MaxQDA (VERBI Software, Marburg, Germany) or NVivo software. In some cases, interviews may be conducted remotely in English.

ELIGIBILITY:
Study participants will be primary school students of schools selected to be included in this study. Schools were selected based on accessibility for the study teams, not having a water source directly connected to the building of the school, and having ≤ 7000 students. 50 students between the ages of 10-12 years old from one or two classes (depending on the number of students in classes) of the 5th-7th grades will be included in the study from each included school. However, due to the large size of the schools and the high number of classes in Nigeria, the 50 students will be selected from two classes of the 5th-7th grades close to where the handwashing stations (Gravit'eau) will be positioned. The 50 selected students will be targeted with the handwashing observation (Module 2) and followed for their hygiene-related health outcomes and absenteeism during the course of the study (Module 4), while 25 of them will be targeted with RANAS and well-being survey (Module 1) and 12 of them will be targeted with collecting their hand-rinse samples (Module 3). Students in the selected classes in each school will be delivered a survey to be self-reported by one of their parents about contextual factors that could affect the hygiene practice of students (Module 5 in Palestine only).

Inclusion criteria Modules 1-4: students must fulfil all the inclusion criteria:

* Primary school students aged 10-12 years attending included schools
* Students must be in the same school for the course of the study (1 year).

Inclusion criteria Module 5: students must fulfil all the inclusion criteria:

- Students of the classes included in the study in each included school in Palestine

Inclusion criteria Module 6:

* Students of the intervention schools
* Students need to represent each included class in the intervention.

The teachers invited to participate in the FGDs should be

* Aged ≥ 18 years old
* Permanent employees in the school
* Teaching one of the classes included in the intervention

Inclusion criteria Module 7:

* The participant needs to be:

  1. a stakeholder within the community, state, or region of the intervention whose position is related in any way to WASH in schools
  2. working in one of the intervention schools. They can be hygiene technicians, teachers, school's principal, or in a leading position in the school.
  3. Aged ≥ 18 years old

     5.3 Exclusion criteria Exclusion criteria Modules 1-4: included students must not fulfil any of the following exclusion criteria:
* Refusal to participate by not providing signed consent and assent forms
* Having any medical condition that prevents them from washing their hands
* Having unexplained intermittent attendance in school (school teachers will be consulted and the school's absenteeism records will be checked for that)
* Not being at the same school for the course of the study (1 year)

Exclusion criteria Module 5: Refusal to participate by the student or his/her parents.

Exclusion criteria Module 6: Refusals to participate.

Exclusion criteria Module 7: Refusals to participate

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2600 (Actual)
Dates: Start 2023-06-29 (Actual); Primary Completion 2024-06-26 (Actual); Study Completion 2024-08-16 (Actual)

PRIMARY OUTCOMES:
Number of participants who wash their hands with water and soap before eating in the school | Up to 12 months
  The primary outcome of the study aims to assess the occurrence, frequency, and technique of participants' handwashing practice with water and soap before eating in the school. This assessment will be conducted through structured observations taking place over a 3-hour period on a single day.

SECONDARY OUTCOMES:
Number of participants who wash their hands with water and soap after using the toilet in the school | Up to 12 months
  The participants' handwashing practice with water and soap after using the toilet in the school will be assessed through structured observations conducted over a single day within a 3-hour period. The observations will focus on capturing the occurrence, frequency, and technique of handwashing.
Change in self-reported handwashing practice | Up to 12 months
  Within the RANAS survey, participants' handwashing practice is assessed using two key event-based inquiries: before eating and after using the toilet. Participants are invited to express their frequency of handwashing on a five-point Likert scale, spanning from "almost never" to "almost always", with "almost always" signifying the most desirable outcome.
Change in self-reported well-being | Up to 12 months
  The well-being of the participants will be evaluated using the KINDL tool which is a questionnaire specifically designed to measure the health-related quality of life in children and adolescents. This questionnaire assesses 6 domains of well-being, including physical health, general feeling, self-feeling, family, friends and school. Participants will respond to the questionnaire using a 5-point Likert scale, which ranges from "almost never" to "almost always". The optimal response, either "almost always" or "almost never," is question-dependent. The domain-specific and overall well-being can be assessed.
Change in the log-transformed number of total coliforms and E.coli CFUs on the hands of participants | Up to 12 months
  Bacterial contamination on the participants' hands will be assessed by quantifying the colony-forming units (CFUs) of E. coli and total coliforms in a sample obtained from their hand rinse. The CFUs will be normalized and transformed using a logarithmic base 10 (log10) to facilitate analysis and comparison
The cumulative count of school absences attributed to hygiene-related illnesses | Up to 8 months
  The daily absenteeism of participants in each cluster, along with the reasons for their absence, will be recorded by a designated teacher. The focus will be on identifying absenteeism incidences due to hygiene-related illnesses such as diarrhoea, respiratory tract infections, helminth infections, head lice, trachoma, and skin infections. The feasibility of these health outcomes will be reassessed with local experts prior to the intervention. To account for the cluster design effect, rates of hygiene-related absenteeism will be calculated separately for each school. This will involve dividing the total number of hygiene-related absences by the number of student-weeks, multiplying the result by 100, and presenting it using descriptive statistics.
The cumulative count of diarrhoea incidences | Up to 8 months
  The cumulative occurrences of diarrhoea, reported during students' absentee tracking by the appointed teacher, will be calculated. To adjust for the cluster design effect, individual school diarrhoea rates will be determined by dividing total instances of diarrhoea by student-weeks, then multiplying the outcome by 100. These rates will be presented using descriptive statistics.
The cumulative count of respiratory tract infections incidences | Up to 8 months
  The cumulative occurrences of respiratory tract infections, reported during students' absentee tracking by the appointed teacher, will be calculated. To adjust for the cluster design effect, individual school diarrhoea rates will be determined by dividing total instances of diarrhoea by student-weeks, then multiplying the outcome by 100. These rates will be presented using descriptive statistics.
The total number of helminth infections incidences | Up to 8 months
  The cumulative occurrences of helminth infections, reported during students' absentee tracking by the appointed teacher, will be calculated. To adjust for the cluster design effect, individual school diarrhoea rates will be determined by dividing total instances of diarrhoea by student-weeks, then multiplying the outcome by 100. These rates will be presented using descriptive statistics.
The total number of head lice incidences | Up to 8 months
  The cumulative occurrences of head lice infections, reported during students' absentee tracking by the appointed teacher, will be calculated. To adjust for the cluster design effect, individual school diarrhoea rates will be determined by dividing total instances of diarrhoea by student-weeks, then multiplying the outcome by 100. These rates will be presented using descriptive statistics.
The total number of trachoma incidences | Up to 8 months
  The cumulative occurrences of trachoma infections, reported during students' absentee tracking by the appointed teacher, will be calculated. To adjust for the cluster design effect, individual school diarrhoea rates will be determined by dividing total instances of diarrhoea by student-weeks, then multiplying the outcome by 100. These rates will be presented using descriptive statistics.
The total number of skin infections incidences | Up to 8 months
  The cumulative occurrences of skin infections, reported during students' absentee tracking by the appointed teacher, will be calculated. To adjust for the cluster design effect, individual school diarrhoea rates will be determined by dividing total instances of diarrhoea by student-weeks, then multiplying the outcome by 100. These rates will be presented using descriptive statistics.

OTHER OUTCOMES:
Covariate 1: Age | Up to 12 months
  Age assessed in years serves as a covariate when estimating the total effect of RANAS factors on handwashing. It will be assessed as part of the combined RANAS and well-being questionnaire, offering answer options within the 10-12 years range.
Covariate 2: Education | Up to 12 months
  Education level serves as a covariate when estimating the total effect of RANAS factors on handwashing. It will be assessed as part of the combined RANAS and well-being questionnaire, providing answer options that span from the third to the seventh grade.
Covariate 3: Sex | Up to 12 months
  Sex serves as a covariate when estimating the total effect of RANAS factors on handwashing. It will be assessed as part of the combined RANAS and well-being questionnaire with two response options: male and female
Covariate 4: Socio-economic status | Up to 12 months
  Socio-economic status serves as a covariate when estimating the total effect of RANAS factors on handwashing. Since directly inquiring about family income from children aged 10-12 years is both difficult and culturally inappropriate, the number of siblings is used as an indicator of the family's socio-economic status. This also provides a proxy for the level of parental attention and hygiene supervision each child might receive, given the number of children the parents have to look after. The information will be collected through the combined RANAS and well-being questionnaire, leaving the response open to the actual number of siblings.
Covariate 5: School water infrastructure | Up to 12 months
  The school infrastructure serves as a covariate when estimating the total effect of RANAS factors on handwashing. This will be assessed through assessing the perceived sufficiency and safety of the school's water supply, satisfaction with the school's available infrastructure for handwashing and obstacles to water access in school. This measure will be part of the combined RANAS and well-being questionnaire offering a five-point Likert scale answers ranging between "Almost never" to "Almost always", with "almost always" signifying the most desirable outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Mirko S. Winler, Prof., Principal Investigator — wiss Tropical and Public Health Institute and University of Basel
Locations (2):
- 26 Primary Schools, Maiduguri, Borno State, Nigeria
- 26 Primary Schools, Hebron, Palestinian Territories

IPD SHARING:
Plan to Share IPD: Yes
The consortium members can share coded or anonymized individual participant data (IPD) internally under the following conditions:
  The ownership of research results belongs to the consortium member(s) whose personnel generated them.
  Each consortium member has the right to utilize the research results of other consortium members for research purposes.
  Research results generated jointly are equally owned by the involved consortium members and can be utilized by all members.
  The use of data by third parties requires written approval from all consortium members.
  After the project is officially concluded and the data has been published, all consortium members are free to conduct secondary data analysis, provided it adheres to ethical agreements and proper acknowledgment is given to the original data.
Supporting Information: Study Protocol
Time Frame: Our partners in Nigeria (Tdh) and Palestine (Cesvi) have direct access to the individual participant data (IPD) as they collect and perform quality control on the data in the field. Other consortium members can request access to the IPD once the data collection is complete and it has been cleaned.
Access Criteria: Within the consortium:
  Data gathered using ODK or KoboToolbox is stored on the ODK central server. The data collecting organizations (Tdh, CESVI), RANAS, and Swiss TPH have direct access to this server. Consortium members who require access to the data can contact someone with server access to request the coded data.
  Outside the consortium:
  Written approval from all consortium members is necessary for third parties to use the data.

REFERENCES:
- [Derived] Galli A, Ma'ani Abuzahra Y, Banziger C, Ballo A, Friedrich MND, Gross K, Harter M, Hattendorf J, Peter M, Tamas A, Owen BN, Winkler MS. Assessing the Effectiveness of a Multicomponent Intervention on Hand Hygiene and Well-Being in Primary Health Care Centers and Schools Lacking Functional Water Supply in Protracted Conflict Settings: Protocol for a Cluster Randomized Controlled Trial. JMIR Res Protoc. 2024 Apr 3;13:e52959. doi: 10.2196/52959. PMID 38569182
- See also: Hands4health project website — http://hands4health.dev/
- See also: Gravit'eau handwashing system website — http://www.graviteau.ch/
- See also: RANAS Ltd. website — http://www.ranasmosler.com/ranas

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-02): https://cdn.clinicaltrials.gov/large-docs/78/NCT05964478/Prot_SAP_000.pdf